CLINICAL TRIAL: NCT06611800
Title: Personalized Advance Prescriptions in Palliative Care at HOME: Interests and Difficulties of Its Implementation (PAPHOME)
Brief Title: Personalized Advance Prescriptions in Palliative Care at HOME: Interests and Difficulties of Its Implementation
Acronym: PAPHOME
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier William Morey - Chalon sur Saône (Other)
Responsible Party: Principal Investigator, Julie COLLOT, Doctor, Centre Hospitalier William Morey - Chalon sur Saône
Other Study IDs: PAPHOME
Record Dates: First submitted 2024-06-11; First posted 2024-09-25 (Actual); Last update posted 2024-10-17 (Actual); Status verified 2024-10

CONDITIONS: Palliative Care

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Presence or absence of personalized advance prescriptions: collection of data for the purpose of know the benefit of personalized advance prescriptions for patients in palliative care at home, particularly in reducing the number of visits to the emergency room and their conditions of death

SUMMARY:
Retrospective data collection on the files of patients cared for by the mobile palliative care team of the William Morey Hospital Center who died in 2022.

DETAILED DESCRIPTION:
Retrospective selection of patients and collection of data : pathology, identified risk, presence of caregiver, end-of-life wishes, characteristics of palliative care treatment, circumstances of death. Comparison of two groups : presence or absence of personalized advance prescriptions.

ELIGIBILITY:
Inclusion Criteria:

* Minimum 18 years old
* Taken care of once in their place of life by a palliative care team
* Died between 01/01/2022 and 12/31/2022 in William Morey Hospital Center

Exclusion Criteria: none

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients over the age of 18 cared for by the mobile palliative care team at the William Morey Hospital Center in Chalon sur Saône, who died between 01/01/2022 and 12/31/2022, having been cared for at least once in their place of life (home, EHPAD) with a visit or a call to the attending physician for advice
Sampling Method: Non-Probability Sample
Enrollment: 256 (Actual)
Dates: Start 2024-10-01 (Actual); Primary Completion 2024-10-01 (Actual); Study Completion 2024-10-07 (Actual)

PRIMARY OUTCOMES:
Know if the presence of advance prescriptions can lead to a reduction in the number of emergency admissions for an "avoidable reason" by its management by a mobile palliative care team (with a maximum of 6 months before death) | A year
  Collection of corresponding variables : presence/absence advance prescriptions ; number of emergency admissions for an "avoidable reason"

SECONDARY OUTCOMES:
Reduction in the number of emergency admissions for all reasons in their last 6 months of life. | A year
  Collection of corresponding variables
Describe conditions of death: location, respect for the wishes of a death at home and notion of a calm death collected from the family | A year
  Collection of corresponding variables
Describe the treatments used for PAPs: Analgesics, Anxiolytics, Anti-secretory drugs, Neuroleptics, Anti-histamines, Anti-emetics | A year
  Collection of corresponding variables

CONTACTS AND LOCATIONS:
Overall Officials: Julie COLLOT, Principal Investigator — Centre Hospitalier William Morey
Locations (1):
- CH William Morey, Chalon-sur-Saône, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Temel JS, Greer JA, Muzikansky A, Gallagher ER, Admane S, Jackson VA, Dahlin CM, Blinderman CD, Jacobsen J, Pirl WF, Billings JA, Lynch TJ. Early palliative care for patients with metastatic non-small-cell lung cancer. N Engl J Med. 2010 Aug 19;363(8):733-42. doi: 10.1056/NEJMoa1000678. PMID 20818875
- [Result] Haun MW, Estel S, Rucker G, Friederich HC, Villalobos M, Thomas M, Hartmann M. Early palliative care for adults with advanced cancer. Cochrane Database Syst Rev. 2017 Jun 12;6(6):CD011129. doi: 10.1002/14651858.CD011129.pub2. PMID 28603881